CLINICAL TRIAL: NCT03044249
Title: Tolerability, Pharmacokinetics, and Efficacy of MP-101 in the Treatment of Patients With Dementia-Related Psychosis and/or Agitation and Aggression
Brief Title: A Study of MP-101 in Dementia-Related Psychosis and/or Agitation and Aggression
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Statistical futility; totality of evidence suggests study unlikely to meet endpoint
Sponsor: Mediti Pharma Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-101-01
Record Dates: First submitted 2017-01-31; First posted 2017-02-06 (Estimated); Results first posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Psychosis; Dementia; Aggression; Agitation; Alzheimer Dementia
Keywords: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders; Dementia; Aggression; Psychomotor Agitation; Alzheimer Disease | interventions — LY2812223

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MP-101 (Experimental): Week 0:
  Participants received 20 milligrams (mg) MP-101 orally QD (1 x 20-mg caps) and 2 placebo caps.
  Week 1:
  Participants received 40 mg MP-101 orally QD (2 x 20-mg caps) and 1 placebo caps.
  Week 2 through Week 9:
  Participants received 60 mg MP-101 orally QD (3 x 20-mg caps ).
  Interventions: Drug: MP-101
- Placebo (Placebo Comparator): Participants received 3 capsules (caps) of placebo orally once daily (QD) during Week 0, Week 1, and Week 2 through Week 9.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MP-101 — Capsules
  Other Names: LY2979165; LY2812223
  Arms: MP-101
Drug: Placebo — Capsules
  Arms: Placebo

SUMMARY:
A ten-week study to assess MP-101 in Dementia-Related Psychosis and/or Agitation and Aggression

ELIGIBILITY:
Inclusion Criteria:

* Females must be of non-childbearing potential, defined as women greater than or equal to (≥) 60 years of age, postmenopausal women ≥50 and less than (<) 60 years of age who have had a cessation of menses for at least 12 months, or women who are congenitally or surgically sterile
* Males must agree to use 2 forms of highly effective birth control with female partners of childbearing potential while enrolled in the study, and for at least 28 days following the last dose
* Ambulatory (with or without walking device) with a stable gait
* Have a Mini-Mental State Examination (MMSE) score of 10 to 24
* Meet clinical criteria for one of the following disorders: dementia associated with Parkinson's disease, dementia with Lewy bodies, possible or probable Alzheimer's disease, frontotemporal degeneration spectrum disorders, vascular dementia
* Able to communicate verbally
* Have an NPI score of ≥4 on either individual item (delusions or hallucinations) or ≥6 on the Psychosis Subscale (combined delusions and hallucinations), or an NPI score of ≥4 on agitation/aggression domain
* Have a reliable caregiver who provides written informed consent to participate and who is in frequent contact with the patient (defined as spending at least 4 hours/day at least 4 days/week with the patient and who is knowledgeable about the patient's daytime and nighttime behaviors). The caregiver must be able to communicate with site personnel, and opinion of the investigator, must understand the written protocol-specified questionnaires. If a caregiver cannot continue, one replacement caregiver will be allowed if the above criterion is met
* Must be on a stable dose of cholinesterase inhibitor and/or memantine, if applicable
* If taking antipsychotic drugs or any drug intended to treat psychosis, must be on a stable treatment regimen for ≥1 month prior to the study
* Have venous access sufficient to allow for blood sampling per the protocol
* Have clinical laboratory test results within normal reference range for the population or investigative site
* Are capable of participating in all study assessments
* Are able and willing to provide consent (patients and caregivers)

Exclusion Criteria:

* Have a history of significant psychotic disorders (including, schizophrenia, delusional disorder, substance abuse psychosis that lasted over 6 months, major depressive disorder or bipolar disorder with psychotic episodes)
* Has a history of ischemic stroke within the last 12 months or any evidence of hemorrhagic stroke
* Have renal impairment as defined by Estimated Glomerular Filtration Rate (eGFR) <45 milliliters per minute per 1.73 square meters (ml/min/1.73m2)
* Have significant cardiovascular, respiratory, gastrointestinal, renal, hematologic, or oncologic comorbidities that could impact patient safety and study participation over 10 weeks
* Have a history of seizures or other condition that would place the patient at increased risk of seizures.
* Are, in the investigator's judgment, at risk for suicide, or as indicated by the Columbia Suicide Severity Rating Scale (C-SSRS)
* Have a Fridericia's corrected QT interval (QTcF) greater than (>) 450 milliseconds (ms) for males or 470 ms for females
* Are currently enrolled in any other clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated, within the last 30 days, in a clinical trial involving an investigational product. If the previous investigational product has a long half-life, at least 3 months (or more) must have passed
* In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mediti Pharma, Study Director — Mediti Pharma Inc.
Locations (20):
- United States (17):
  - Dignity Health (St. Joseph Hospital and Medical Center), Phoenix, Arizona
  - Neuro-Therapeutics Inc, Pasadena, California
  - Associated Neurologists of Southern CT, Fairfield, Connecticut
  - Marcus Neuroscience Institute, Boca Raton, Florida
  - Meridien Research, Brooksville, Florida
  - Galiz Research, Hialeah, Florida
  - Galiz Research, Miami Springs, Florida
  - CNS, Orlando, Florida
  - Parkinson's Disease Treatment Center of SW Florida, Port Charlotte, Florida
  - Meridien Research Inc, St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - College Park Family Care Neuro, Overland Park, Kansas
  - J. Gary Booker, MD, Clinical Trials, Shreveport, Louisiana
  - Alzheimer's Research Corporation, Paterson, New Jersey
  - Clarity Clinical Research, East Syracuse, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Neurology Diagnostics Inc, Dayton, Ohio
- Canada (3):
  - SKDS Research Inc., Newmarket, Ontario
  - Montreal Neurological Institute, Montreal, Quebec
  - Centre de recherche sur le vieillissement du CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | MP-101
Started | 42 | 39
Received at Least One Dose of Study Drug | 42 | 39
Completed | 32 | 25
Not Completed | 10 | 14
Not completed — Adverse Event | 4 | 9
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-compliance with Study Drug | 1 | 0
Not completed — Study Terminated by Sponsor | 2 | 0
Not completed — Withdrawal by Subject | 2 | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- MP-101: Week 0:
  Participants received 20 mg MP-101 orally QD (1 x 20-mg caps) and 2 placebo caps.
  Week 1:
  Participants received 40 mg MP-101 orally QD (2 x 20-mg caps) and 1 placebo caps.
  Week 2 through Week 9:
  Participants received 60 mg MP-101 orally QD (3 x 20-mg caps ).
- Total: Total of all reporting groups
Arm/Group | Placebo | MP-101 | Total
Number analyzed (Participants) | 42 | 39 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (9.44) | 74.0 (7.66) | 74.7 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 30 | 33 | 63
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 37 | 34 | 71
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 2 | 3 | 5
  United States | 40 | 36 | 76
Neuropsychiatric Inventory (NPI) Psychosis Score [Mean (Standard Deviation); unit: units on a scale] — The NPI Psychosis subscale score was the sum of the delusions and hallucinations items of the standard 12-item NPI that measured psychosis symptoms in participants with dementia. Scores for each subscale (frequency x severity) were calculated for each item score and ranged from 0 to 24 with higher scores indicating more frequent and/or severe neuropsychiatric symptoms.
  units on a scale | 8.4 (6.36) | 7.7 (5.70) | 8.0 (6.02)
NPI Agitation/Aggression Score [Mean (Standard Deviation); unit: units on a scale] — The NPI Psychosis subscale score for Agitation/Aggression consists of Agitation/Aggression item of the standard 12-item NPI that measured psychosis symptoms in participants with dementia. Scores for each subscale (frequency x severity) were calculated for each item score and ranged from 0 to 12 with higher scores indicating more frequent and/or severe neuropsychiatric symptoms.
  units on a scale | 5.8 (3.34) | 5.3 (3.15) | 5.5 (3.24)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 30% Improvement From Baseline in the Neuropsychiatric Inventory (NPI) - Psychosis Subscale or Aggression/Agitation Subscale Score
Description: The NPI is a questionnaire that quantifies behavioral changes in dementia. For each of 12 domains there are 4 scores: Frequency (scale:1=occasionally to 4=very frequently), Severity (scale:1=Mild to 3=Severe), Total (frequency x severity), Caregiver distress (scale: 0=not at all distressing to 5=extremely distressing). An NPI response was defined as at least a 30% improvement from baseline on the NPI Psychosis sub-score (for participants with a psychosis diagnosis (Delusions and Hallucinations)) or the NPI Aggression/Agitation sub-score (for participants with an agitation/aggression diagnosis). The delusions, hallucinations, and aggression/agitation domain scores were added together to form a core total score with score range of 0 to 36. Lower score=less severity. A negative change score from baseline indicates improvement.
Time Frame: Week 10
Population: All randomized participants who received at least one dose of study drug who completed at least Week 4 with NPI scores but were not withdrawn due to early termination of the study.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received 3 capsules of placebo orally once daily (QD) during Week 0, Week 1 and Week 2 through Week 9.
- MP-101: Week 0:
  Participants received 20 mg MP-101 orally QD ((1 x 20-mg caps and 2 placebo caps)).
  Week 1:
  Participants received 40 mg MP-101 orally QD ((2 x 20-mg caps and 1 placebo caps)).
  Week 2 through Week 9:
  Participants received 60 mg MP-101 orally QD (3 x 20-mg caps ).
Arm/Group | Placebo | MP-101
Number analyzed (Participants) | 33 | 26
percentage of participants | 58 | 62
Statistical Analysis 1: Comparison: Placebo vs MP-101; Test type: Superiority; p = 0.48, Fisher Exact; Response Ratio = 4, 90% CI 2-sided [-18 to 25]

2. Secondary Outcome: Percentage of Participants With Improvement From Baseline in the Clinical Global Impression of Improvement (CGI-I) at Week 10
Description: The CGI rating scale, which measures symptom severity, treatment response and the efficacy of treatments, is used in clinical studies on mental disorders. CGI Improvement scale is a 7 point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Time Frame: Week 10
Population: All randomized participants who received at least one dose of study drug who had a baseline and at least one post-baseline CGI-I measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | MP-101
Number analyzed (Participants) | 32 | 25
percentage of participants
  Very much improved | 0 | 8.0
  Much improved | 25.0 | 28.0
  Minimally improved | 34.4 | 28.0
  No change | 21.9 | 16.0
  Minimally worse | 15.6 | 12.0
  Much worse | 3.1 | 8.0
  Very much worse | 0 | 0

3. Secondary Outcome: Change From Baseline in NPI Total Score
Description: The NPI is a questionnaire that quantifies behavioral changes in dementia. For each of 12 domains there are 4 scores: Frequency (scale: 1=occasionally to 4=very frequently), Severity (scale:1=Mild to 3=Severe), Total (frequency x severity), Caregiver distress (scale: 0=not at all distressing to 5=extremely distressing). The NPI Total Score is calculated by adding the Individual Item Scores for all 12 domains, to yield a possible NPI Total Score of 0 to 144. Lower score=less severity. A negative change score from baseline indicates improvement.
Time Frame: Baseline, Week 10
Population: All randomized participants who received at least one dose of study drug who completed at least Week 4 with NPI scores.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | MP-101
Number analyzed (Participants) | 34 | 26
score on a scale | -3.43 (2.34) | -8.70 (2.66)
Statistical Analysis 1: Comparison: Placebo vs MP-101; Test type: Superiority; p = 0.14, Mixed Models Analysis; Mean Difference (Final Values) = -5.28, 90% CI 2-sided [-11.16 to 0.61]

4. Secondary Outcome: Change From Baseline in NPI Core Total Score
Description: The NPI is a questionnaire that quantifies behavioral changes in dementia. For each of 12 behavioral domains there are 4 scores: Frequency (scale: 1=occasionally to 4=very frequently), Severity (scale:1=Mild to 3=Severe), Total (frequency x severity), Caregiver distress (scale: 0=not at all distressing to 5=extremely distressing). The NPI CoreTotal Score is calculated by adding the Individual Item Scores for all 3 domains (hallucinations, delusions, and agitation/aggression) to yield a possible NPI Core Total Score of 0 to 36. Lower score=less severity. A negative change score from baseline indicates improvement.
Time Frame: Baseline, Week 10
Population: All randomized participants who received at least one dose of study drug who completed at least Week 4 with NPI scores.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | MP-101
Number analyzed (Participants) | 34 | 26
score on a scale | -3.46 (1.15) | -5.05 (1.31)
Statistical Analysis 1: Comparison: Placebo vs MP-101; Test type: Superiority; p = 0.37, Mixed Models Analysis; Mean Difference (Final Values) = -1.58, 90% CI 2-sided [-4.47 to 1.31]

5. Secondary Outcome: Number of Participants With NPI Caregiver Distress
Description: The NPI is a questionnaire that quantifies behavioral changes in dementia. For each of 12 domains there are 4 scores: Frequency (scale:1=occasionally to 4=very frequently), Severity (scale:1=Mild to 3=Severe), Total (frequency x severity), Caregiver distress (scale:0=not at all distressing to 5=extremely distressing). The NPI Psychosis Subscale Caregiver Distress Score is calculated by adding Individual Item Scores for the domains of Delusions and Hallucinations, to yield a possible total score of 0 to 10. Lower score=less severity. A negative change score from baseline=improvement.
Time Frame: Week 10
Population: All randomized participants who received at least one dose of study drug who completed at least Week 4 with NPI scores.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MP-101
Number analyzed (Participants) | 34 | 26
Participants
  Week 10 Delusions ( Not at all) | 0 | 0
  Week 10 Delusions ( Minimally) | 1 | 1
  Week 10 Delusions (Mildly) | 9 | 5
  Week 10 Delusions (Moderately) | 7 | 3
  Week 10 Delusions (severely) | 1 | 2
  Week 10 Delusions (Very Severely or extremely) | 1 | 0
  Week 10 Hallucinations ( Not at all) | 3 | 1
  Week 10 Hallucinations ( Minimally) | 3 | 3
  Week 10 Hallucinations (Mildly) | 3 | 4
  Week 10 Hallucinations (Moderately) | 6 | 2
  Week 10 Hallucinations (severely) | 1 | 1
  Week 10 Hallucinations (Very Severely or extremely) | 0 | 0

6. Secondary Outcome: Change From Baseline in NPI Domains - Anxiety
Description: The 12 individual items in NPI that quantify changes in dementia are delusions, hallucinations, agitation, depression, anxiety, apathy, disinhibition, irritability, euphoria, aberrant motor behavior, nighttime behaviors, and appetite. For each of 12 behavioral domains there are 4 scores: Frequency (scale:1=occasionally to 4=very frequently), Severity (scale:1=Mild to 3=Severe), Total (frequency x severity), Caregiver distress (scale: 0=not at all distressing to 5=extremely distressing). The NPI Psychosis Subscale Anxiety consists of anxiety item to yield a possible NPI Score of 0 to 12. Lower score=less severity. A negative change score from baseline indicates improvement.
Time Frame: Baseline, 10 Weeks
Population: All randomized participants who received at least one dose of study drug who completed at least Week 4 with NPI scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | MP-101
Number analyzed (Participants) | 32 | 25
units on a scale | -0.1 (3.53) | -0.6 (2.69)

7. Secondary Outcome: Number of Participants With Any Treatment Emergent Adverse Event
Description: Number of participants with untoward medical occurrences that emerge during the treatment period, having been absent pretreatment, or worsen relative to the pretreatment state, which do not necessarily have a causal relationship with this treatment. A summary of serious adverse events (SAEs) and other non-serious adverse events (AEs) is located in the reported adverse events module.
Time Frame: Baseline Up to 10 Weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MP-101
Number analyzed (Participants) | 42 | 39
Participants | 24 | 24

8. Secondary Outcome: Change From Baseline in the Unified Parkinson's Disease Rating Scale (UPDRS) Part III
Description: Part III of the UPDRS is an investigator-scored scale used to assess the motor symptoms of patients with Parkinson's disease. The investigator rates the patient on 14 items based on observation or the performance of a task the patient performs (even in the context of any comorbidities) on a 5-point scale. The scores range from 0 to 4, with higher scores indicating greater impairment. The total UPDRS score was calculated as the sum of all items, ranging from 0 to 56 with higher scores indicating greater impairment. If any individual item was missing, the UPDRS score was be set to missing.
Time Frame: Baseline, Week 10
Population: All randomized participants who received at least one dose of study drug who completed at least Week 4 with NPI scores.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MP-101
Number analyzed (Participants) | 34 | 26
units on a scale | -0.29 (0.76) | -0.37 (0.87)
Statistical Analysis 1: Comparison: Placebo vs MP-101; Test type: Superiority; p = 0.94, Mixed Models Analysis; Mean Difference (Final Values) = -0.08, 90% CI 2-sided [-2.00 to 1.84]

9. Secondary Outcome: Population Pharmacokinetics (PK): Plasma Levels of MP-101 and Metabolite
Description: Summary statistics of sparse blood concentration samples at weeks 2, 4, 6, 10 and Early Termination obtained utilizing a population PK approach.
Time Frame: Week 2: 4-8 hours post-dose; Week 4: Predose, 0-2 hours postdose; Week 6: 8-12 hours postdose; Week 10: 2- 4 hours;Early Termination
Population: All participants who received at least one dose of MP-101 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomoles per liter (nmol/L)
Groups:
- MP-101; LY2812223 (MP-101 Metabolite): Participants received 60 mg MP-101 orally QD (3 x 20-mg caps).
Arm/Group | MP-101 | LY2812223 (MP-101 Metabolite)
Number analyzed (Participants) | 34 | 34
Nanomoles per liter (nmol/L)
  Week 2: 4-8 hours: number analyzed (Participants) | 17 | 25
  Week 2: 4-8 hours | 7.9 (1.11) | 429.8 (1.00)
  Week 4: Predose: number analyzed (Participants) | 0 | 22
  Week 4: Predose |  | 85.0 (1.01)
  Week 4: 0-2 hours: number analyzed (Participants) | 14 | 25
  Week 4: 0-2 hours | 11.4 (1.09) | 249 (1.01)
  Week 6: 8-12 hours: number analyzed (Participants) | 11 | 22
  Week 6: 8-12 hours | 4.1 (1.36) | 808.4 (1.00)
  Week 10: 2- 4 hours: number analyzed (Participants) | 16 | 20
  Week 10: 2- 4 hours | 9.3 (1.12) | 929 (1.00)
  Early Termination: number analyzed (Participants) | 1 | 4
  Early Termination | NA (NA) — For N=1, individual value 1 was reported. | 13.0 (1.24)

ADVERSE EVENTS:
Time Frame: Baseline Up To 10 Weeks
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Placebo | MP-101
All-Cause Mortality (participants affected / at risk) | 0/42 | 1/39
Serious Adverse Events (participants affected / at risk) | 4/42 | 4/39
Other Adverse Events (participants affected / at risk) | 12/42 | 22/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | MP-101 (N=39)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Unresponsive to stimuli (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | MP-101 (N=39)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Fatigue (General disorders) | 2 (2) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 3 (4)
Dizziness (Nervous system disorders) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 2 (2) | 5 (5)

LIMITATIONS AND CAVEATS:
Statistical futility; totality of evidence suggests study unlikely to meet endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/49/NCT03044249/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03044249/SAP_001.pdf